CLINICAL TRIAL: NCT05242263
Title: Reducing Attention Bias Variability Using Attention Control Training With Feedback Among Individuals With Posttraumatic Stress Disorder
Brief Title: ACT With Feedback for Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor Yair Bar-Haim, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAU-ABV
Record Dates: First submitted 2022-01-27; First posted 2022-02-16 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: PTSD
Keywords: PTSD; Attention Training; Cognitive Bias Modification; Attention Bias Modification
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either active or sham feedback in a 1:1 ratio.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Study design is a double-blind parallel-group RCT: two groups (ACT+feedback and ACT+sham feedback), and three assessment time points (pre-, post-treatment and follow up). The independent clinical evaluators, personnel staff who deliver the training, and participants are blind before and during treatment to group allocation, which is coded with a random number for each condition. Participants are randomly assigned to conditions in a 1:1 ratio using a list created with a random number generator. The random assignment list was created before enrollment to the study started. Group assignment is monitored by a staff member not involved in the study in any other capacity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group - ACT with feedback (Experimental): At the beginning of each session participants will complete 45 standard dot-probe trials. During these trials, participants' ABV will be measured and set as their baseline. In the following trials, participants will receive feedback: a green screen background when their ABV will reach below their baseline or a red screen background when their baseline ABV score is surpassed.
  Interventions: Behavioral: Attention Control Training (ACT) with ABV feedback
- Control group - ABV with yoked sham feedback (Sham Comparator): Participants in this group will receive sham feedback that is unrelated to their ABV during the task, this is by presenting a feedback given to another participant in the training group (i.e., yoked sham feedback).
  Interventions: Behavioral: Attention Control Training (ACT) with yoked sham feedback

INTERVENTIONS:
Behavioral: Attention Control Training (ACT) with ABV feedback — At the beginning of each session, participants will complete 45 standard dot-probe trials as described above. Participants' ABV on these trials will be calculated and set as their personal baseline (see below for ABV calculation). In the following 165-training trials, participants will receive feedback: when their online-calculated ABV will be below their baseline screen background will be green whereas its color will be red when their online ABV score will be higher than their baseline. Patients will be instructed to try to keep the background green for as long as possible.
  Arms: Training group - ACT with feedback
Behavioral: Attention Control Training (ACT) with yoked sham feedback — Participants in this group will be exposed to the same task as in the active group but will receive sham feedback that is unrelated to their ABV during task performance. They will be presented with a feedback that is yoked to the one given to a participant in the training group.
  Arms: Control group - ABV with yoked sham feedback

SUMMARY:
The purpose of this study is to explore the efficacy of Attention Control Training with the inclusion of feedback for Post Traumatic Stress Disorder (PTSD).

It seems that the most efficient ABMT method to balance attention bias variability (ABV) among individuals with PTSD is Attention Control Training (ACT). This type of training is designed to balance attention allocation towards threat-related and neutral stimuli. A few studies have further shown that this training type succeeds in balancing the aberrant fluctuations in attention bias observed in patients with PTSD, and that this leads to a reduction in PTSD symptoms (Badura-Brack et al., 2015).

The purpose of the current study is to examine the efficacy of ACT that also includes feedback. Specifically, we intend to test whether the inclusion of feedback on top of standard ACT may enhance training efficacy in reducing ABV and in reducing PTSD symptoms.

DETAILED DESCRIPTION:
The aim of the current study is to explore the efficacy of Attention Control Training with the inclusion of feedback for Post Traumatic Stress Disorder (PTSD).

Individuals with PTSD exhibit increased threat-related attention bias variability (ABV; Lacoviello et al., 2014; Naim et al., 2015). Based on these findings, computerized training methods aimed to modify the attention bias were developed (Attention Bias Modification Training; ABMT).

It seems that the most efficient ABMT method to balance ABV among individuals with PTSD is Attention Control Training (ACT). This type of training is designed to balance attention allocation towards threat-related and neutral stimuli. A few studies have further shown that this training type succeeds in balancing the aberrant fluctuations in attention bias observed in PTSD, and that this leads to a reduction in PTSD symptoms (Badura-Brack et al., 2015).

The purpose of the current study is to examine the efficacy of ACT that also includes a feedback component. Specifically, we intend to test whether the inclusion of feedback on top of standard ACT may enhance training efficacy in reducing ABV and in reducing PTSD symptoms.

For this purpose, we will recruit 60 IDF veterans diagnosed with PTSD that will be randomly assigned to one of two conditions: ACT with feedback or ACT with yoked sham feedback.

We expect that ACT with feedback will produce greater reduction in PTSD symptoms and in ABV relative to ACT with yoked sham feedback.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD according to the DSM-5 and related to military service, ages 18-65

Exclusion Criteria:

* Psychotic or Bipolar disorder, drug and alcohol abuse, other psychological treatment, vision problems that are not overcome with regular glasses, physical disability that prevents ability to operate computer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the total severity score of the CAPS-5 interview | Measurements at Baseline, 1 week post treatment, and 3-months follow-up post treatment
  The Clinician Administered PTSD Scale (CAPS-5), is a structured interview that will be used to make a diagnosis of PTSD according to the DSM-V criteria. This interview is consists of 30 items regarding the frequency and intensity of PTSD symptoms and a total score of severity is been rated, with higher scores denoting higher symptom severity.

SECONDARY OUTCOMES:
Change from baseline of the total score of the PTSD Checklist (PCL-5) | Measurements at Baseline, 1 week post treatment, and 3-months follow-up post treatment
  The PCL-5, is a 20-item National Center for PTSD Checklist of the Department of Veterans Affairs. Scores can range from 0 to 80, with higher scores reflecting more symptoms of PTSD.
Change from baseline of the total score of the PHQ-9 | Measurements at Baseline, 1 week post treatment, and 3-months follow-up post treatment
  The PHQ-9 is a 9-item scale for depression symptoms (Kroenke, Spitzer, & Williams, 2001). Scores can range from 0 to 27, with higher scores reflecting more symptoms of depression.

OTHER OUTCOMES:
Post-Training Attention Bias Variability | Measurements at Baseline, 1 week post treatment, and 3-months follow-up post treatment
  Change in Attention Bias Variability from Baseline to Post-training measurement and follow-up. ABV is calculated in four steps: 1) a trial-by trial moving average algorithm computed reaction times for all successive 10 neutral trial blocks and all successive 10 threat trial blocks, 2) successive attention bias scores were calculated by subtracting the first threat block average from the first neutral block average, the second threat block average from the second neutral block average, etc., forming a series of consecutive attention bias scores, 3) the standard deviation of these successive bias scores was then calculated, providing an index of variation in attention bias throughout the session, and 4) this standard deviation score was divided by the participant's mean overall reaction time
The Credibility/Expectancy Questionnaire (CEQ) | Measurements at Baseline, 1 week post treatment, and 3-months follow-up post treatment
  The Credibility/Expectancy Questionnaire (CEQ; Devilly & Borkovec, 2000). This instrument consists of 6 items which derive two factors: expectancy for change and treatment credibility. This CEQ will be used to explore whether expectancies or treatment credibility are related to outcomes.
The CGI-I | 1 week post treatment, and 3-months follow-up post treatment
  Severity and improvement scale (CGI-I) will be used to assess participants global clinical condition. The CGI-I is single-item, clinician-reported, measure assessing severity and improvement of illness using a 7-point Likert-type scale.
The CGI-S | 1 week post treatment, and 3-months follow-up post treatment
  Severity and improvement scales (CGI-S ) will be used to assess participants global clinical condition. The CGI-S is single-item, clinician-reported, measure assessing severity and improvement of illness using a 7-point Likert-type scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naim R, Abend R, Wald I, Eldar S, Levi O, Fruchter E, Ginat K, Halpern P, Sipos ML, Adler AB, Bliese PD, Quartana PJ, Pine DS, Bar-Haim Y. Threat-Related Attention Bias Variability and Posttraumatic Stress. Am J Psychiatry. 2015 Dec;172(12):1242-50. doi: 10.1176/appi.ajp.2015.14121579. Epub 2015 Jul 24. PMID 26206076
- [Background] Badura-Brack AS, Naim R, Ryan TJ, Levy O, Abend R, Khanna MM, McDermott TJ, Pine DS, Bar-Haim Y. Effect of Attention Training on Attention Bias Variability and PTSD Symptoms: Randomized Controlled Trials in Israeli and U.S. Combat Veterans. Am J Psychiatry. 2015 Dec;172(12):1233-41. doi: 10.1176/appi.ajp.2015.14121578. Epub 2015 Jul 24. PMID 26206075